CLINICAL TRIAL: NCT05955209
Title: An Open, Single Arm, Single Center Phase II Clinical Study Evaluating the Efficacy and Safety of RC48-ADC in the Treatment of Metastatic Castration Resistant Prostate Cancer (mCRPC) Progression After Novel Endocrine Therapy
Brief Title: Clinical Study on the Efficacy and Safety of RC48-ADC in the Treatment of Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDTYPEC053
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: RC48-ADC; metastasis Castration Resistant Prostate Cancer; HER2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin(RC48-ADC) (Experimental): Disitamab Vedotin(RC48-ADC) :2.0mg/kg，Q2W
  Interventions: Drug: Disitamab Vedotin（RC48-ADC）

INTERVENTIONS:
Drug: Disitamab Vedotin（RC48-ADC） — Participants will receive RC48-ADC intravenous injection (2.0 mg/kg, Q2W) until disease progression or death.
  Other Names: RC48

SUMMARY:
This is a single-arm, open, single-center clinical study to evaluate the efficacy and safety of RC48-ADC in patients with mCRPC who have progressed after NHT. A total of 40 patients with mCRPC with immunohistochemically confirmed HER2 expression who had progressed after treatment with at least one novel endocrine therapy will be included in this study.

DETAILED DESCRIPTION:
This is a single-arm, open, single-center clinical study to evaluate the efficacy and safety of RC48-ADC in patients with mCRPC who have progressed after NHT. A total of 40 patients with mCRPC with immunohistochemically confirmed HER2 expression who had progressed after treatment with at least one novel endocrine therapy will be included in this study. Participants will receive RC48-ADC intravenous injection (2.0 mg/kg, Q2W) until disease progression or death. During the treatment, participants will evaluate every 4 weeks, including PSA testing every 4 weeks and tumor evaluation according to PCWG3 standards every 8 weeks. If the patient develops disease progression, the treatment will be discontinued and survival follow-up will be conducted every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) Prostate cancer confirmed by histology;
* 2) ≥ 18 years old;
* 3) The presence of metastatic lesions confirmed by bone scan and/or CT/MRI and/or PET-CT;
* 4) ECOG score 0-2;
* 5) Continuously maintain ADT treatment and maintain testosterone levels ≤ 50ng/dL; The progression of prostate cancer recorded within 6 months prior to screening;
* 6) Having received at least one NHT in the past before progressing;
* 7) HER2 IHC 1+, 2+, or 3+;
* 8) Inability to or refusal docetaxel chemotherapy;
* 9) Voluntarily join the study;
* 10) Expected survival time ≥ 6 months;
* 11) Normal function of main organs;

Exclusion Criteria:

* 1)Have a history of malignant tumors other than prostate cancer;
* 2)Previously received allogeneic stem cell or parenchymal organ transplantation;
* 3) Previously or currently suffering from congenital or acquired immunodeficiency diseases;
* 4) The patient have a history of allergy to RC48 or paclitaxel, or a history of Hypersensitivity to chimeric or humanized antibodies or fusion proteins, or allergy to excipients of the study drug;
* 5) Other significant clinical and laboratory abnormalities that affect safety evaluation;
* 6) Those who are unwilling or unable to take effective contraceptive measures;
* 7) Subjects with active brain metastasis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
PSA response rate | 24 months
  The proportion of subjects receiving at least one cycle of treatment with the study drug who had at least a 50% reduction in PSA from baseline and maintained it for more than 21 days (PSA50).

SECONDARY OUTCOMES:
ORR，Objective Response Rate | 24 months
  The proportion of patients who achieved patial response and complete reponse.
Overall survival (OS) | From the first dose to death from any cause，up to two years.
  median OS or OS rate
Progression free survival | From the first dose to the first documentation of disease progression or death, up to two years.
  median PFS or PFS rate

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: Yes
Article publication
Supporting Information: Study Protocol
Time Frame: Determine after article publication
Access Criteria: Determine after article publication